CLINICAL TRIAL: NCT00489151
Title: A Randomized Study Comparing Lamivudine Versus Adefovir Dipivoxil for Prevention of zHBV Reactivation in HBsAg Seropositive Patients Undergoing Cytotoxic Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 04-315 T/637; HARECCTR0500002
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Hepatitis B
Keywords: HBV
MeSH Terms: conditions — Hepatitis B | interventions — adefovir dipivoxil; Lamivudine

INTERVENTIONS:
Drug: adefovir dipivoxil
Drug: lamivudine

SUMMARY:
Liver diseases due to hepatitis B reactivation are serious causes of morbidity and mortality in hepatitis B infected patients treated with chemotherapy. We have previously shown that with pre-emptive use of lamivudine, one can drastically reduce liver-related morbidity and mortality in such patients. However, due to the development of hepatitis B virus resistance to lamivudine, some of these hepatitis B infected patients still develop hepatitis. This is a research study aiming to compare the use of adefovir dipivoxil to lamivudine in hepatitis B infected patients treated with chemotherapy. Both of these drugs have been approved for the treatment of the hepatitis B infection in the United States, European Union and Hong Kong.

All patients who were recruited in this study will receive study medication, either lamivudine 100 mg daily or adefovir dipivoxil 10 mg daily to cover the entire period of chemotherapy for 72 weeks. All patients will be follow-up for an additional 24 weeks thereafter. Altogether, 70 subjects will be recruited from Queen Mary Hospital, Hong Kong SAR.

This is an open-label study, which means that the patients and the study doctor will know which treatment the subjects are assigned into. If a subject decides to take part in the study and is found eligible, he/she will be randomly (like flipping of coin) assigned to one of the following dose groups:

Lamivudine (100 mg) tablet Adefovir dipivoxil (10 mg) tablet

ELIGIBILITY:
Inclusion Criteria:

* HBsAg+, nucleoside/nucleotide analogue naïve, malignant disease for iv chemotherapy

Exclusion Criteria:

* HCV+ HDV+

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-06; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
To compare the development of viral resistance to anti-viral therapy: lamivudine versus adefovir dipivoxil in immunosuppressed patients | 72 weeks

SECONDARY OUTCOMES:
To assess the safety of adefovir dipivoxil in HBV seropositive patients who are planned to undergo chemotherapy, as compared to lamivudine. | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, Dr, Principal Investigator — Department of Medicine, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, Hong Kong, China